CLINICAL TRIAL: NCT00556387
Title: Possible Neuroprotective Effects of Ketamine in Children With Severe Traumatic Brain Injury
Brief Title: Efficacy of Ketamine in Children With Severe Brain Injury for Brain Cell Protection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been withdraw from the IRB. The PI has transferred to another university. The IND was transferred.
Sponsor: University of Arkansas (Other)
Responsible Party: Carole Hamon, Regulatory Affairs Manager, University of Arkansas for Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 86674; 86674
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo Group receiving Saline Infusion.
  Interventions: Drug: saline
- 2 (Experimental): Case Group receiving Ketamine infusion.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: saline — 1 mg/kg IV bolus slowly over 1-2 minutes followed by 0.5 mg/kg IV continuous infusion over 48 hours or until discontinuation of ICP monitor (whichever occurs first)
  Arms: 1
Drug: Ketamine — 1 mg/kg IV bolus slowly over 1-2 minutes, followed by 0.5 mg/kg IV continuous infusion for 48 hours or until discontinuation of ICP monitor (whichever occurs first)
  Arms: 2

SUMMARY:
The purpose of this study is to determine the possible effects of an anesthetic agent called Ketamine on the injured brain in children.

The researchers think that it will effect the outcomes of children with these injuries.

ELIGIBILITY:
Inclusion Criteria:

* are 1 month to 16 years of age; AND
* are admitted to the PICU following severe TBI (any GCS 3-8 inclusive) within 8 hours after the injury; AND
* are intubated and ventilated for the management of TBI; AND
* are anticipated to have an indwelling arterial or venous catheter for blood sampling during the first three days of study enrollment; AND
* have an intra-cranial pressure (ICP) monitoring device for management of TBI.

Exclusion Criteria:

* are less than 4 kilograms in weight upon admission
* are less than 1 month of age;
* are greater than 16 years of age;
* have a clinical diagnosis of non-accidental TBI;
* have suffered immersion injury or prolonged hypoxic injury (lasting greater than 10 minutes);
* have a known allergy to ketamine;
* have a planned removal of endotracheal tube or the removal of central venous catheter AND arterial catheter within 72 hours of study enrollment;
* have a current history of neuromuscular disease;
* have a current history of hepatic failure;
* have a current history of glaucoma
* require chronic treatment with anti-epileptic drugs (AEDs) or devices;
* more than 8 hours have elapsed from the time of injury to PICU admission;
* have documentation of a positive pregnancy test at the time of enrollment;
* if there is a lack of commitment to aggressive intensive care therapies (the subject is either on a DNR status due to pre-existing medical condition, or the family decides to withdraw support prior to participation in the study due to other multiple severe injuries and organ failures resulting from the trauma).

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To compare clinical, radiological, and neurodevelopmental outcomes between children who receive ketamine vs placebo infusions following traumatic brain injury. | 1 year

SECONDARY OUTCOMES:
To compare the expression of biomarkers of CNS injury between cases and controls. | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Muayyad Tailounie, MD, Principal Investigator — Arkansas Children's Hospital Research Institute